CLINICAL TRIAL: NCT04913506
Title: Evaluation of the Effects of Neuromuscular Electrical Stimulation and Mirror Therapy in Hemiplegia Rehabilitation; Prospective, Randomized, Controlled, Single-Blinded Study
Brief Title: Evaluation of the Effects of Neuromuscular Electrical Stimulation and Mirror Therapy in Hemiplegia Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Burcu Metin Ökmen, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BYIEAH-H
Record Dates: First submitted 2021-05-26; First posted 2021-06-04 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Hemiplegia; Upper Extremity Dysfunction
Keywords: hemiplegia; mirror theraphy; NMES
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Controlled, Single-Blinded Study
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Mirror (Active Comparator): Along with conventional rehabilitation techniques, patients will be given ROM exercises in all directions, in front of the real mirror, by the practitioner on the healthy upper extremity for 30 minutes.
  Interventions: Other: Group Mirror
- Group NMES (Active Comparator): Along with conventional rehabilitation techniques, NMES will be applied to the hemiplegic arm for 30 minutes by the practitioner while the patients are sitting in a chair.
  Interventions: Device: Group NMES
- Group Mirror+NMES (Active Comparator): In addition to conventional rehabilitation techniques, patients will be given ROM exercises for 30 minutes in all directions in front of the real mirror to the healthy extremity, which the practitioner will synchronize with visual or auditory stimuli, and NMES treatment for 30 minutes to the paretic upper extremity.
  Interventions: Other: Group Mirror+NMES

INTERVENTIONS:
Other: Group Mirror — For 30 minutes, ROM exercises will be applied to the solid upper extremity in all directions in front of a real mirror by the practitioner. (3 weeks, 5 days a week, 15 sessions in total)
  Other Names: Mirror theraphy
  Arms: Group Mirror
Device: Group NMES — NMES will be applied to the hemiplegic arm(deltoid, elbow extensors and forearm) for 30 minutes by the practitioner (3 weeks, 5 days a week, 15 sessions in total)
  Other Names: NMES (neuromuscular electrical stimulation)
  Arms: Group NMES
Other: Group Mirror+NMES — The practitioner will be synchronized with visual or auditory stimuli, and ROM exercises in all directions in front of the real mirror for 30 minutes, and NMES therapy for 30 minutes on the paretic upper extremity will be applied together. (3 weeks, 5 days a week, 15 sessions in total)
  Other Names: Mirror therapy+NMES
  Arms: Group Mirror+NMES

SUMMARY:
In this study, it was aimed to evaluate whether or not NMES in front of the mirror brings an additional benefit to mirror therapy alone or NMES alone on upper extremity motor and functional development, spasticity, anxiety, depression, cognitive function and activities of daily living, and neuropathic pain.

DETAILED DESCRIPTION:
Cerebrovascular diseases are the general name given to clinical neurological pictures that occur as a result of pathological changes in the blood vessels of the primary lesion and / or in the properties of the blood passing through them. Many complications develop in the acute and chronic periods in patients with stroke, and the rate of complication development has been reported to vary between 40-96% in different studies. The aim of hemiplegic upper extremity rehabilitation is to prevent complications and improve lost motor-sensory control. Upper limb rehabilitation is less successful than lower limb rehabilitation because the upper limb is more functional and more complex.

For muscle reeducation, NMES is used to strengthen inhibited muscle groups, facilitate voluntary isolated muscle contraction, prevent muscle atrophy, increase metabolism and enzyme activity, change the contractile properties of the muscle, maintain or increase the normal range of motion of the joint, develop voluntary movement and functional gains. NMES has been used in hemiplegia rehabilitation since 1960 for the purpose of functional retraining of muscles. The purpose of this treatment is to enable the muscles with impaired neural function of the electrical current to perform a functional and useful movement.

Applications in front of the mirror are thought to trigger the neuronal connections in the motor cortex associated with the imagined movement. Findings obtained from studies with functional magnetic resonance support this theory. Compared to conventional PR, applications in front of the mirror are thought to have more and longer-lasting effects.

ELIGIBILITY:
Inclusion Criteria:

* Subacute hemiplegia
* Patients who can communicate well, are motivated enough and are willing to participate in the study
* Patients' medical conditions are stable
* Initiation of voluntary extension movement in the wrist (lower limit)

Exclusion Criteria:

* The presence of more than one previous cerebrovascular disease (except transient ischemic attack).
* Presence of flaccid hemiplegia.
* Presence of a previous neurological disease causing a decrease in strength in the affected extremity.
* Presence of deformity due to a previous fracture, inflammatory arthropathy, etc. in the affected extremity.
* Presence of more than grade 3 spasticity in upper extremity according to Modified Ashworth Scale
* Use of cardiac pace maker
* Presence of fatal cardiac arrhythmia
* Presence of seizure history within 2 years.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Extremity Motor Rating Scale | Change from Baseline Fugl-Meyer Upper Extremity Motor Rating Scale at 3rd week
  To analysis the increase in upper limb motor function Motor score: ranges from 0 (hemiplegia) to 100 points (normal motor performance). Divided into 66 points for upper extremity and 34 points for the lower extremity. Sensation: ranges from 0 to 24 points. Divided into 8 points for light touch and 16 points for position sense.

SECONDARY OUTCOMES:
Mini-Mental Test | Change from Baseline Mini-Mental Test at 3rd week
  for cognitive functions
Numeric Rating Scale | Change from Baseline Numeric Rating Scale at 3rd week
  for pain
Pain Detect Questionnaire | Change from Baseline Pain Detect Questionnaire at 3rd week
  for neuropathic pain
Functional Independence Scale (FIM) | Change from Baseline Functional Independence Scale (FIM) at 3rd week
  for daily life activities
Modified Tardieu Scale | Change from Baseline Modified Tardieu Scale at 3rd week
  Score, Description 0, No resistance during movement.
  1. There is very slight resistance during movement, but no noticeable "catch".
  2. There is a noticeable "catch" at a certain angle, followed by relaxation.
  3. Clonus occurring at a certain angle and lasting for seconds (ending with fatigue).
  4. Uninterrupted clonus occurring at a certain angle and lasting for more than 10 seconds. 5, The joint is too stiff to move (petrified).
Brunnstrom stages | Change from Baseline Brunnstrom stages at 3rd week
  For improvement of upper limb motor function

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Metin Ökmen, M.D. Assoc. Prof, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital; Büşra Yeşil, M.D., Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- Bursa Yüksek İhtisas Eğitim ve Araştırma Hastanesi, Bursa, Turkey (Türkiye)